CLINICAL TRIAL: NCT01003795
Title: P-REWARDS (Promus - Registry Experience at the Washington Hospital Center, DES)
Brief Title: Promus - Registry Experience at the Washington Hospital Center, Drug-eluting Stent (DES)
Acronym: P-REWARDS
Status: Withdrawn | Type: Observational
Why Stopped: Not Funded
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: P REWARDS
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Promus: Patients treated with at least one Promus, everolimus-eluting, Stent

SUMMARY:
Single-center registry of patients treated with at least one Promus, everolimus-eluting, Stent, with the primary objective to assess clinical success and safety at 30 days, 6 months and 1 year post-implantation.

DETAILED DESCRIPTION:
Interventional cardiology was revolutionized by the invention of stents, initially with the bare-metal stents (BMS) and recently with the drug-eluting stents (DES). The everolimus eluting stents have shown very promising results in randomized clinical trials, demonstrating a reduction of clinical and angiographic restenosis in comparison to BMS, and comparable clinically-driven target lesion revascularization rates in comparison with sirolimus-eluting stents. While registry data is available from outside of the United States, it will be important to collect "real-world" data regarding the stent usage and outcomes in the United States. In this study we propose to follow patients who received at least one Promus® Stent for at least 1 year post initial stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, >18 years of age
* Patients who received at least one Promus drug-eluting stent at the Washington Hospital Center

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with at least one Promus, everolimus-eluting, Stent at the Washington Hospital Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Major Adverse Cardiac Events (MACE) post Promus Stent implantation | Follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Research Institute/Cardiovascular Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States